CLINICAL TRIAL: NCT04905953
Title: Comparison Of Different Doses Of Intrathecal Neostigmine In Prevention Of Post-Dural Puncture Headache: Prospective, Randomized, Controlled, Triple-blinded Trial
Brief Title: Comparison Of Different Doses Of Intrathecal Neostigmine In Prevention Of Post-Dural Puncture Headache
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Fathy, Lecturer of anesthesia and SICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N-128-2020
Record Dates: First submitted 2021-03-16; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Neostigmine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Neostigmine — Intrathecal injection of two doses of neostigmine (10 & 20 mic) during spinal anesthesia for cesarean section.

SUMMARY:
We hypothesized that; intrathecal administration of neostgmine in spinal anesthesia may have a beneficial role in reduction of the incidence or severity of PDPH.

DETAILED DESCRIPTION:
Neostigmine will be administered in two different doses (10 & 20 mic) in addition to 10mg bupivicaine intrathecally for cesarean section compared to control group where 10 mg bupivicaine in addition to 20mic fentanyl will be administered intrathecally. The primary outcome will be detection of the incidence of postdural puncture headache (PDPH). A 25-gauge Quincke spinal needle will be used for spinal anesthesia.Patients indicated for elective caesarean section surgery will be included in the study. The exclusion criteria are contraindications for regional anesthesia including local infection, hemorrhagic disorders, drug hypersensitivity, muscular disorders and central and peripheral neuropathy, and drug abuse history and addiction.

Other outcomes will include age, ASA class, and duration of surgery. Sensory and motor function will be assessed every minute until T4 level is reached. Hemodynamic status (systolic and diastolic blood pressures, heart rate, and SPO2) will be recorded every 3 minutes throughout the surgery and then 4 hourly thereafter, for 24 h postoperatively. Recovery time from spinal anesthesia (return of motor power of both lower limbs) will be also recorded by anesthesiologist who is unaware of the group. Also the intra-operative and recovery phase complications including nausea, vomiting, itching, dyspnea, respiratory rate less than 10 per min, hypoxia (SPO2 less than 92% on room air), bradycardia (HR less than 60bpm), and hypotension (SPB less than 90) will be recorded.

Postoperative assessment will include pain scores "Overall 24-h VAS score", recorded at 30-min interval for first 4 h and then 4 hourly thereafter, for 24 h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for elective caesarean section surgery

Exclusion Criteria:

* Contraindications for regional anesthesia including local infection, hemorrhagic disorders, drug hypersensitivity, muscular disorders and central and peripheral neuropathy, and drug abuse history and addiction.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females candidate for elective cesarean section
Enrollment: 274 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of PDPH following spinal anesthesia for cesarean section surgery. | 72 hours.
  Diagnosis of PDPH is as follows, it is severe and described as "searing and spreading like hot metal," involving the back and front of the head, and spreading to the neck and shoulders, sometimes involving neck stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelaal Ahmed Mahmoud A, Mansour AZ, Yassin HM, Hussein HA, Kamal AM, Elayashy M, Elemady MF, Elkady HW, Mahmoud HE, Cusack B, Hosny H, Abdelhaq M. Addition of Neostigmine and Atropine to Conventional Management of Postdural Puncture Headache: A Randomized Controlled Trial. Anesth Analg. 2018 Dec;127(6):1434-1439. doi: 10.1213/ANE.0000000000003734. PMID 30169405